CLINICAL TRIAL: NCT04465240
Title: Adolescent Responses to Varying Environments in Virtual Reality Simulations (THRIVE: The Research In Virtual Environments Study)
Brief Title: Adolescent Responses to Varying Environments in Virtual Reality Simulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Daniel Hackman, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 262625; 1R21HD099596-01 (NIH); UP-19-00205 (Other: University of Southern California)
Record Dates: First submitted 2020-06-11; First posted 2020-07-10 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Residential Characteristics; Emotions; Stress, Psychological; Stress, Physiological
Keywords: Neighborhoods; Poverty Areas; Adolescent Development
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality simulation of neighborhood disadvantage (Experimental): Participants will attend one study session. They will watch a video during a baseline rest period. Participants will be assigned to navigate and explore the virtual neighborhood representative of disadvantage they were assigned to. Then they will watch a video again during a recovery period.
  Interventions: Other: Virtual reality
- Virtual reality simulation of neighborhood affluence (Active Comparator): Participants will attend one study session. They will watch a video during a baseline rest period. Participants will be assigned to navigate and explore the virtual neighborhood, representative of affluence they were assigned to. Then they will watch a video again during a recovery period.
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — Participants are immersed in a neighborhood environment in virtual reality

SUMMARY:
The objective of this study, named THRIVE (The Research In Virtual Environments Study), is to test hypotheses for how neighborhood environments influence stress and emotion, as a mechanism by which they may influence health. Neighborhood environments may have both acute influences on stress-related processes, but also may have lifespan effects due to the chronic, cumulative effects of repeated exposures and the long-term toll of adapting to adverse neighborhood environments. However, assessing neighborhood influences on stress and emotion is methodologically challenging. This study develops such a novel, alternative approach to address these questions by deploying a virtual reality (VR) based model of neighborhood disadvantage and affluence that creates an immersive experience approximating the experience of being in different neighborhoods. In this study, this model will be applied to understand neighborhood effects in a diverse sample of adolescents (n = 130) from a range of disadvantaged and affluent neighborhoods. The proposed study will employ a randomized experiment (n = 65 per condition), with online questionnaires and a single study session, to determine (a) if virtual exposure to neighborhood disadvantage elicits differences in emotion and stress reactivity; (2) if growing up in a disadvantaged neighborhood results in habituation or sensitization to different neighborhood characteristics; and (3) if chronic stress results in habituation or sensitization to different neighborhood characteristics. This research will develop an innovative methodology that will help establish the role that neighborhoods may play in eliciting stress as well as the processes of adaptation to chronic stress and chronic neighborhood exposures. In addition, it will help establish a method that can be utilized more broadly to study contextual and social environmental influences on psychological and biological risk in adolescence.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Are able to use a dominant hand for joystick manipulation and a non- dominant hand for physiological measurements,
* Are in good physical and mental health, with no self-reported history of hypertension, cardiovascular disease (CVD) or CVD treatment (with associated medication list indicative of treatments that result in exclusion),
* Have hair at least 1cm in length based on self-report to be able to provide a hair sample.

Exclusion Criteria:

* Pregnant, by self-report

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Hackman, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California / USC Suzanne Dworak-Peck School of Social Work, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 107 participants were enrolled, eight withdrew after enrollment but prior to randomization to condition, without attending the single study session. Thus while enrollment was 107 the total started in the protocol flow was 99.
Groups:
- Virtual Reality Simulation of Neighborhood Disadvantage: Participants will attend one study session. They will watch a video during a baseline rest period. Participants will be assigned to navigate and explore the virtual neighborhood representative of disadvantage they were assigned to. Then they will complete questionnaires and watch a video again during a recovery period.
  Virtual reality: Participants are immersed in a neighborhood environment in virtual reality
- Virtual Reality Simulation of Neighborhood Affluence: Participants will attend one study session. They will watch a video during a baseline rest period. Participants will be assigned to navigate and explore the virtual neighborhood, representative of affluence they were assigned to. Then they will complete questionnaires and watch a video again during a recovery period.
  Virtual reality: Participants are immersed in a neighborhood environment in virtual reality
Period: Overall Study
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Started | 50 | 49
Completed | 50 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.03 (1.06) | 15.85 (1.16) | 15.94 (1.11)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 20 | 16 | 36
    Male | 30 | 33 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American / Black | 3 | 2 | 5
  Asian | 6 | 5 | 11
  Latinx / Hispanic | 21 | 19 | 40
  Multiracial | 6 | 4 | 10
  Native American, American Indian or Alaskan Native | 0 | 2 | 2
  Other | 1 | 0 | 1
  White | 13 | 17 | 30
Parental Education [Count of Participants; unit: Participants] — Highest level of education attained by a parent/caregiver
  Participants
    High School Education or Less | 5 | 4 | 9
    Some College or Associate's Degree | 7 | 2 | 9
    Bachelor's Degree | 20 | 21 | 41
    Master's Degree | 13 | 16 | 29
    Doctoral Degree or Equivalent | 5 | 6 | 11
Neighborhood Poverty Rate [Mean (Standard Deviation); unit: % below poverty in neighborhood] — For each participant, this represents the percentage of families with incomes below the poverty line in the U.S. census tract (neighborhood) that the participant resides within. Based on American Communities Survey five- year estimates from 2015-2019. Population: One address could not be accurately geocoded and assigned a U.S. census tract, leading to one fewer participant for this baseline measure
  % below poverty in neighborhood
    number analyzed (Participants) | 50 | 48 | 98
    (all) | 11.56 (11.02) | 9.82 (8.3) | 10.71 (9.77)

OUTCOME MEASURES:

1. Primary Outcome: Emotional Response
Description: Multiple measures were used for emotion felt in the VR neighborhood:
  1. Participants rate how strongly they felt 9 specific emotions (0-8 scale; 0 indicates none, 8 is the strongest possible feeling).
  2. Two composite scores based on averaging responses for specific emotions: Positive emotion (enthusiasm, contentment, amusement) and Negative emotion (fear, sadness, disgust, anger). Averages were based on the standard score representing standard deviations above/below the mean. The mean score was 0. Positive emotion ranged from -1.9, the lowest positive emotion, to 2.0, the highest. Negative emotion ranged from -0.7, the lowest negative emotion, to 3.5, the highest. A positive score reflects greater than average for that type of emotion, and negative score reflects less than average for that type of emotion.
  3. Self-Assessment Manikin (SAM) scale: two dimensional scales for how they felt, from (a) happy to unhappy (1 to 9), and (b) excited to calm (1 to 9) (Bradley & Lang, 1994)
Time Frame: Immediately after the virtual reality task (average of 28 minutes post baseline)
Population: Two participants (one from each arm) were excluded from analyses due to major technical problems / glitches in virtual reality presentation that lead to invalid data. One participant did not complete the measure of happy/unhappy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Number analyzed (Participants) | 49 | 48
units on a scale
  Amusement: from 0 (not at all) to 8 (strongest ever felt) | 3.65 (1.82) | 4.31 (1.75)
  Anger: from 0 (not at all) to 8 (strongest ever felt) | 1.29 (1.89) | 0.33 (0.81)
  Contentment / Happiness: from 0 (not at all) to 8 (strongest ever felt) | 2.98 (1.65) | 4.54 (1.88)
  Compassion: from 0 (not at all) to 8 (strongest ever felt) | 3.18 (2.09) | 2.56 (2.32)
  Disgust: from 0 (not at all) to 8 (strongest ever felt) | 2.86 (2.42) | 0.69 (1.36)
  Enthusiasm/excitement: from 0 (not at all) to 8 (strongest ever felt) | 2.69 (1.97) | 3.77 (2.21)
  Fear: from 0 (not at all) to 8 (strongest ever felt) | 1.59 (2.21) | 0.44 (0.92)
  Sadness: from 0 (not at all) to 8 (strongest ever felt) | 2.67 (2.37) | 0.33 (0.69)
  Surprise: from 0 (not at all) to 8 (strongest ever felt) | 2.84 (2.31) | 2.79 (2.62)
  Positive Emotion: Composite based on enthusiasm, contentment, amusement (Overall mean is 0) | -0.28 (0.76) | 0.28 (0.91)
  Negative Emotion: Composite based on fear, sadness, disgust, anger (Overall mean is 0) | 0.41 (0.98) | -0.42 (0.34)
  Happy-Unhappy: from 1 (happy) to 9 (unhappy) [Self-Assessment Manikin (SAM)] | 4.58 (1.66) | 3.4 (1.61)
  Excited-calm: from 1 (excited) to 9 (calm) [Self-Assessment Manikin (SAM)]: number analyzed (Participants) | 48 | 48
  Excited-calm: from 1 (excited) to 9 (calm) [Self-Assessment Manikin (SAM)] | 5.39 (1.96) | 5.85 (1.98)

2. Primary Outcome: Salivary Cortisol
Description: Concentration of the stress hormone cortisol in saliva samples, measured in (µg/dL), that participants provide over the course of the study session to assess cortisol response
Time Frame: Measured 5 times: (1) end of baseline, (2) after virtual reality (VR) neighborhood (VR: 11 minutes, average), (3) after questionnaires (26 minutes after VR end, average), (4) video (recovery), after first 15 minutes, (5) after final 15 minutes of video
Population: Two participants (one from each arm) were excluded from analyses due to major technical problems / glitches in virtual reality that lead to invalid data. Sixteen participants (7 in virtual affluent condition, 9 in virtual disadvantaged condition) were removed due potential contamination between saliva samples across time in the study session.
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Number analyzed (Participants) | 40 | 41
µg/dL
  Baseline (end) | 0.121 (0.063) | 0.135 (0.123)
  Virtual Reality Neighborhood (immediately after) | 0.134 (0.066) | 0.182 (0.156)
  Questionnaire completion | 0.251 (0.333) | 0.287 (0.395)
  Video, After 15 minutes | 0.261 (0.419) | 0.361 (0.584)
  Video, After 30 minutes | 0.279 (0.542) | 0.286 (0.473)

3. Primary Outcome: Blood Pressure
Description: Systolic (SBP) and diastolic (DBP) blood pressure, in mmHG, measured and summarized across epochs in the study session.
Time Frame: Measured in 5 epochs, typical 60-90 minutes total: (1) Baseline before virtual reality (VR), (2) VR neighborhood (11 minutes, average), (3) Questionnaires (begins 6 minutes after VR end, average), (4) Video: first 15 minutes, (5) Video, final 15 minutes
Population: Two participants (one from each arm) were excluded from analyses due to major technical problems / glitches in virtual reality that lead to invalid data. One participant did not have blood pressure recordings and for one technical problems led to data not being recorded.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Number analyzed (Participants) | 47 | 48
mmHG
  SBP, Baseline (mean, in mmHg) | 120.45 (17.65) | 117.79 (19.78)
  SBP, VR neighborhood (mean, in mmHg) | 123.82 (23.46) | 125.97 (19.13)
  SBP, Questionnaires (mean, in mmHg) | 120.41 (16.13) | 114.11 (17.46)
  SBP, Video, First 15 Minutes (mean, in mmHg) | 115.29 (20.16) | 113.02 (23.54)
  SBP, Video, Second, 15 Minutes (mean, in mmHg) | 110.90 (22.62) | 113.79 (17.52)
  DBP, Baseline (mean, in mmHg) | 70.14 (13.64) | 66.23 (13.65)
  DBP, VR neighborhood (mean, in mmHg) | 76.29 (15.13) | 72.28 (16.22)
  DBP, Questionnaires (mean, in mmHg) | 69.18 (11.91) | 68.22 (14.35)
  DBP, Video, First 15 Minutes (mean, in mmHg) | 70.50 (15.91) | 67.31 (17.29)
  DBP, Video, Second 15 Minutes (mean, in mmHg) | 66.07 (13.89) | 67.20 (11.22)

4. Primary Outcome: Respiratory Sinus Arrhythmia (RSA)
Description: Respiratory Sinus Arrhythmia (RSA) reflects parasympathetic nervous systemt activity and is used as an index of emotion regulation, with higher scores indicating greater parasympathetic activation. It is derived from the natural log of the power of high frequency heart rate variability (heart rate variability is the variability in the amount of time in between heart beats, and high frequency heart rate variability is the power of activity in the 0.15-0.4 Hz range). Based on electrocardiograph signals measured and summarized across epochs in the study session.
Time Frame: as for outcome 3
Population: Two participants (one from each arm) were excluded from analyses due to major technical problems / glitches in virtual reality that lead to invalid data. One participant had technical problems led to data not being recorded, and another had minimal signal recorded across data collection.
Measure: Mean (Standard Deviation); unit: ms-squared
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Number analyzed (Participants) | 48 | 47
ms-squared
  RSA, Baseline (Mean) | 6.56 (0.90) | 6.31 (1.12)
  RSA, VR neighborhood (Mean) | 6.88 (0.79) | 6.69 (1.15)
  RSA, Questionnaires (Mean) | 6.77 (0.80) | 6.65 (1.16)
  RSA, Video, First 15 Minutes (Mean) | 6.76 (0.88) | 6.79 (1.04)
  RSA, Video, Second 15 Minutes (Mean) | 6.89 (0.82) | 6.90 (0.90)

5. Primary Outcome: Cardiac Output (CO)
Description: Cardiac Output (CO) represents the volume of blood pumped by the heart (L/min). Increasing values indicate greater volume of blood pumped per unit time. Derived from impedance cardiography signals measured and and then summarized across epochs in the study session.
Time Frame: as for outcome 3
Population: Two participants (one from each arm) were excluded from analyses due to major technical problems / glitches in virtual reality that lead to invalid data. One participant had technical problems led to data not being recorded, and four had minimal or low quality signal recorded across data collection.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Number analyzed (Participants) | 47 | 45
L/min
  CO, Baseline (mean) | 5.35 (1.99) | 5.50 (2.13)
  CO, VR neighborhood (mean) | 5.37 (1.79) | 5.90 (2.42)
  CO, Questionnaires (mean) | 5.18 (1.74) | 5.29 (1.70)
  CO, Video, First 15 Minutes (mean) | 5.30 (1.82) | 5.12 (1.73)
  CO, Video, Second 15 Minutes (mean) | 5.28 (1.72) | 5.15 (1.62)

6. Primary Outcome: Total Peripheral Resistance (TPR)
Description: Total peripheral resistance (TPR) is an index of an index of vasoconstriction (mean arterial pressure divided by cardiac output). Increasing values indicate greater vasoconstriction. Derived from impedance cardiography signals measured and and then summarized across epochs in the study session.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg*min/L
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Number analyzed (Participants) | 47 | 45
mmHg*min/L
  TPR, Baseline (mean) | 18.82 (8.88) | 19.29 (12.80)
  TPR, VR neighborhood (mean) | 19.62 (8.28) | 18.05 (9.19)
  TPR, Questionnaires (mean) | 18.29 (7.55) | 18.04 (10.04)
  TPR, Video, First 15 Minutes (mean) | 19.07 (9.65) | 18.83 (9.79)
  TPR, Video, Second 15 Minutes (mean) | 17.96 (9.21) | 18.88 (9.29)

7. Primary Outcome: Pre-ejection Period (PEP)
Description: Pre-ejection period (PEP) is a measure of sympathetic nervous system activation. Higher values indicate greater sympathetic activation. Derived from impedance cardiography (Q-point in ECG to B-point in impedance cardiography), signals are measured and and then summarized across epochs in the study session.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
Number analyzed (Participants) | 47 | 45
ms
  PEP, Baseline (mean) | 114.69 (7.43) | 117.92 (7.64)
  PEP, VR neighborhood (mean) | 112.49 (6.42) | 113.84 (8.64)
  PEP, Questionnaires (mean) | 112.97 (6.68) | 114.60 (8.68)
  PEP, Video, First 15 Minutes (mean) | 114.29 (6.94) | 115.58 (7.43)
  PEP, Video, Second 15 Minutes (mean) | 113.28 (7.04) | 114.75 (8.18)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the single study session included in the study (up to 4-5 hours)
Arm/Group | Virtual Reality Simulation of Neighborhood Disadvantage | Virtual Reality Simulation of Neighborhood Affluence
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT04465240/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT04465240/SAP_001.pdf
  • Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT04465240/ICF_002.pdf